CLINICAL TRIAL: NCT05503407
Title: Baseline V-RESOLVE Score Guided Versus Angiography Guided Stent Implantation in Coronary Bifurcation Lesions (CIT-RESOLVE II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Kefei Dou, MD, Professor, China National Center for Cardiovascular Diseases
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-1361
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Coronary Bifurcation Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline V-RESOLVE score-guided PCI (Experimental): Lesions with baseline V-RESOLVE <14 scores would undergo either jailed wire technique or provisional two-stent strategy;
  Lesions with baseline V-RESOLVE ≥14 scores would undergo either jailed balloon technique or elective two-stent strategy.
  Interventions: Procedure: Baseline V-RESOLVE score-guided PCI
- Angiography-guided PCI (Placebo Comparator): The choice of interventional strategy was left to the discretion of experienced interventionists based on the coronary angiogram.
  Interventions: Procedure: Angiography-guided PCI

INTERVENTIONS:
Procedure: Baseline V-RESOLVE score-guided PCI — Jailed wire technique (JWT): Both main vessel (MV) and side branch (SB) are wired. The MV is stented with wire protection in SB. If suboptimal results exist, the SB would be rewired and a kissing balloon inflation (KBI) is undertaken.
  Jailed balloon technique: A monorail balloon is advanced into the SB. If there is TIMI flow grade decrease in the SB after MV stenting, the SB balloon is inflated to simulate attempt to reopen the SB.
  Provisional two-stent strategy: Lesion preparation and MV stenting are consistent with JWT. Provisional SB stenting could be undertaken when suboptimal results occur after SB rewiring and a KBI is undertaken.
  Elective two-stent strategy: Patients in this subgroup would undergo crush procedure or any other elective two-stent strategy which usually stenting SB before MV stenting.
  Arms: Baseline V-RESOLVE score-guided PCI
Procedure: Angiography-guided PCI — The choice of interventional strategy was left to the discretion of experienced interventionists based on the coronary angiogram.
  Arms: Angiography-guided PCI

SUMMARY:
The purpose of this study is to investigate whether baseline V-RESOLVE score guided intervention is associated with significant reduction of side branch occlusion rates compared to angiography guided intervention in patients with coronary bifurcation lesions.

DETAILED DESCRIPTION:
A number of 1104 patients scheduled for elective percutaneous coronary intervention (PCI) with native coronary bifurcation lesions suitable for stent implantation are included in the present study. This study will be conducted in two stages with 552 patients each. In the first stage, all patients receive angiography-guided PCI. In the second stage, all patients receive PCI under the guidance of baseline V-RESOLVE score.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Inclusion Criteria:

   1. Subject must be male or nonpregnant female ≥18 years of age and ≤75 years of age;
   2. Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia;
   3. Subject is eligible for PCI;
   4. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed;
   5. Subject is willing to comply with all protocol-required follow-up evaluation.
2. Angiographic Inclusion Criteria:

   1. Subjects have coronary bifurcation lesions requiring PCI with stent implantation according to clinical guidelines and/or the operator's judgement;
   2. Visually estimated reference vessel diameter (RVD) of target main vessel ≥2.5 mm and ≤4.0 mm;
   3. Visually estimated RVD of target side branch ≥ 2.0mm;
   4. Coronary anatomy is likely to allow delivery of a study device to the target lesion(s);

Exclusion Criteria:

1. Clinical Exclusion Criteria:

   1. Subject has a known allergy to contrast (that cannot be adequately pre-medicated) and/or the trial stent system or protocol-required concomitant medications (e.g., stent alloy, stainless steel, sirolimus, everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors, or aspirin);
   2. Planned surgery within 6 months after the index procedure;
   3. Subject has one of the following (as assessed prior to the index procedure):

      * Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 12 months;
      * Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.);
      * Planned procedure that may cause non-compliance with the protocol or confound data interpretation;
   4. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions;
   5. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint;
   6. Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure;
   7. Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure);
   8. Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential);
   9. Subject with left ventricular ejection fraction < 35%;
   10. Subject has preoperative renal dysfunction: serum creatinine>2.0mg/dl (176.82umol/L).
2. Angiographic Exclusion Criteria:

   1. Left main lesions;
   2. In case of acute myocardial infarction of which the culprit vessel located at the left anterior descending (LAD) artery, the bifurcation lesion (LAD/diagonal branch [RVD>2.5mm]) which is proximal to occluded LAD segment should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1104 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
side branch occlusion after main vessel stenting | Immediately after the main vessel
  The primary endpoint is side branch occlusion, which is defined as any decrease in TIMI flow grade or absence of flow in side branch after main vessel stent well opposed.

SECONDARY OUTCOMES:
The elevation of biomarkers of periprocedural myocardial injury [Creatine Kinase-Myocardial Band (CK-MB) and Troponin I]. | 48h after Percutaneous Coronary Intervention (PCI)
  Periprocedural Myocardial Infarction (MI) is defined by the Society for Cardiovascular Angiography and Interventions criteria.
Major adverse cardiac events (MACE) | 12-month follow-up
  Including all cause death, all myocardial infarction (MI) and target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Kefei Dou, MD, PhD, Principal Investigator — Fuwai Hospital and National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China